CLINICAL TRIAL: NCT05594745
Title: Comparative Efficacy of Different Treatment Regimens in Patients With Dry Eye Disease and Meibomian Gland Dysfunction
Brief Title: Treatment Regimens in Meibomian Gland Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tauber Eye Center (Other)
Responsible Party: Principal Investigator, Joseph Tauber, Principal Investigator, Tauber Eye Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TEC_IIR2020
Record Dates: First submitted 2022-10-20; First posted 2022-10-26 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast

STUDY DESIGN:
Intervention Model Description: Multiple group, single unmasked randomized trial
Who Masked: Investigator
Masking Description: Randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Xiidra (Active Comparator): one drop BID for 9 months
  Interventions: Drug: Lifitegrast Ophthalmic; Device: Lipiflow
- Systane (Active Comparator): One drop QID for 9 months
  Interventions: Drug: Systane Free; Device: Lipiflow

INTERVENTIONS:
Drug: Lifitegrast Ophthalmic — eyedrop
  Other Names: Xiidra
  Arms: Xiidra
Drug: Systane Free — eyedrop
  Arms: Systane
Device: Lipiflow — thermal pulsation
  Other Names: thermal pulsation

SUMMARY:
This study seeks to explore the relevance of inflammation in dry eye patients with MGD and compare the efficacy of LipiFlow treatment followed by lid hygiene and lubricant treatment with Systane Ultra or LipiFlow treatment followed by lid hygiene and lifitegrast treatment in patients with meibomian gland dysfunction.

DETAILED DESCRIPTION:
The role of inflammation as a central mechanism of pathophysiology in dry eye disease has been well documented, including both clinical and basic science studies. It has been estimated that 50-75% of patients complaining of dry eyes have meibomian gland dysfunction (MGD). As defined by TFOS DEWs II MGD is a chronic, diffuse abnormality of the meibomian glands, commonly characterized by terminal duct obstruction and/or qualitative/quantitative changes in the glandular secretion. This may result in the alteration of the tear film, symptoms of eye irritation, clinically apparent inflammation, and ocular surface disease. It has been estimated that 86% of patients complaining of dry eye disease demonstrate meibomian gland dysfunction. The role of ocular surface inflammation vs. the role of obstructive meibomian gland disease is less well understood.

The symptoms of MGD (evaporative dry eye) may be difficult to differentiate from those of dry eye syndrome (aqueous deficient dry eye (ADDE)), though MGD patients tend to report more burning and stinging than they report complaints of grittiness, sandiness or foreign body sensation in the eyes. However, there is a significant lack of association between signs and symptoms in patients with dry eye disease, which makes it extremely difficult to sort out which patients would benefit from which treatment options. Given the high prevalence of dry eye in the general population any attempt to segregate patients into appropriate treatment types is important.

Traditional treatment options for MGD include the use of artificial lubricants (some lipid-containing such as Systane Ultra), warm lid compresses using cloths or heat pads of various materials, systemic tetracyclines and episodic treatment with topical antibiotics or antibiotic/steroid combinations. Eyelid thermal pulsation procedures (e.g. LipiFlow) have helped many patients. Only one published study supports the benefit of anti-inflammatory treatment (lifitegrast) in patients with MGD. This study seeks to explore the relevance of inflammation in dry eye patients with MGD and compare the efficacy of LipiFlow treatment followed by lid hygiene and lubricant treatment with Systane Ultra or LipiFlow treatment followed by lid hygiene and lifitegrast treatment in patients with meibomian gland dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18 or older, of any sex and any race. 2. Clinical diagnosis of MGD, defined as:

1. complaints of burning, stinging or dryness > 40 on scale of 0-100.
2. thickened secretions or occlusion of > 4 of eight assessed glands of the central lower eyelid.
3. clinically evident redness of the eyelid margin > 1+ on a scale of 0-4. 4. Willing to comply with the protocol instructions. 5. Has read (or has had read to), understood, and signed an Informed Consent.

   -

   Exclusion Criteria:
   * 1. Active ocular infection or ocular inflammatory disease. 2. Anterior basement membrane dystrophy or history of recurrent erosion syndrome.

     3. History of severe / serious ocular pathology or other medical condition that could result in an inability to safely complete the study. 4. Ocular surgery, LipiFlow or iLux or IPL or MG duct probing within past 6 months.

     5. Participation by the patient in any other investigational study within the past 30 days.

     6. Unlikely to comply with protocol instructions for any reason (confusion, substance abuse, etc.).

   The Principal Investigator or the Medical Monitor reserves the right to declare a patient ineligible based on medical evidence that indicates the patient is unsuitable for the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-01-21 (Actual); Study Completion 2023-01-21 (Actual)

PRIMARY OUTCOMES:
eye dryness score | 9 months
  visual analog scale from 0 to 100, higher is worse

SECONDARY OUTCOMES:
corneal flurescein staining | 9 months
  NEI corneal staining scale scored from 0 to 4, higher is worse
ocular discomfort score | 9 months
  visual analog scale from 0 to 100, higher is worse

CONTACTS AND LOCATIONS:
Locations (1):
- joseph Tauber, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lemp MA, Crews LA, Bron AJ, Foulks GN, Sullivan BD. Distribution of aqueous-deficient and evaporative dry eye in a clinic-based patient cohort: a retrospective study. Cornea. 2012 May;31(5):472-8. doi: 10.1097/ICO.0b013e318225415a. PMID 22378109
- [Background] Nichols KK, Nichols JJ, Mitchell GL. The lack of association between signs and symptoms in patients with dry eye disease. Cornea. 2004 Nov;23(8):762-70. doi: 10.1097/01.ico.0000133997.07144.9e. PMID 15502475
- [Background] Nelson JD, Shimazaki J, Benitez-del-Castillo JM, Craig JP, McCulley JP, Den S, Foulks GN. The international workshop on meibomian gland dysfunction: report of the definition and classification subcommittee. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):1930-7. doi: 10.1167/iovs.10-6997b. Print 2011 Mar. No abstract available. PMID 21450914
- [Background] Starr CE, Gupta PK, Farid M, Beckman KA, Chan CC, Yeu E, Gomes JAP, Ayers BD, Berdahl JP, Holland EJ, Kim T, Mah FS; ASCRS Cornea Clinical Committee. An algorithm for the preoperative diagnosis and treatment of ocular surface disorders. J Cataract Refract Surg. 2019 May;45(5):669-684. doi: 10.1016/j.jcrs.2019.03.023. PMID 31030780